CLINICAL TRIAL: NCT01982903
Title: Prospective Study of Urinary Connective Tissue Growth Factor and Related Pro-fibrotic Mediators as Potential Early Biomarkers of Progressive Renal Allograft Fibrosis in de Novo Kidney Recipients
Brief Title: Prospective Study of Urinary Markers of Fibrosis in Kidney Transplants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr Thomas Vanhove, Dr Thomas Vanhove, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: s55992
Record Dates: First submitted 2013-10-31; First posted 2013-11-13 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Failure
Keywords: kidney transplantation; connective tissue growth factor; fibrosis
MeSH Terms: conditions — Renal Insufficiency; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — whole blood, serum, urine, renal allograft tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney transplant recipients: Adult recipients of a primary or secondary cadaveric or living donor single renal allograft at the University Hospitals Leuven between July 2014 and June 2016

SUMMARY:
The purpose of this study is to determine whether urinary connective tissue growth factor (uCTGF) can predict the onset of fibrosis in transplanted kidneys.

DETAILED DESCRIPTION:
Since March 2004, and as part of routine clinical practice, protocol renal allograft biopsies are routinely performed at implantation and at 3, 12 and 24 months after transplantation, in all patients who receive a kidney transplant at the University Hospitals Leuven, unless there is a medical contra-indication or patient refusal to undergo this procedure. The biopsies are scheduled using a dedicated Microsoft Access database ("Biopsy Database"), that is maintained on the central servers of the University Hospitals Leuven. Patients who have an unexplained change in renal allograft function, undergo additional clinically indicated indication biopsies. These biopsies are also recorded in the aforementioned Microsoft Access Database.

All clinical data, including pretransplant donor and recipient characteristics, and post-transplant follow-up data are directly stored and maintained in a prospectively collected electronic database (CCL database until 06/2012, transferred to the central KWS database in 2012). This electronic database is the only existing clinical database for these patients, and contains all clinical patient charts. No written records are collected.

All renal allograft biopsies will be scored by a single renal pathologist according to the most recent Banff classification, blinded for the clinical parameters and timing of the biopsy. These rescoring data are directly entered in the dedicated Microsoft Access database ("Biopsy Database").

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive a primary or secondary single cadaveric or living donor renal allograft.
* Signed informed consent

Exclusion Criteria:

* Patients receiving a combined renal allograft.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult recipients of a primary or secondary cadaveric or living donor single renal allograft at the University Hospitals Leuven.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Allograft interstitial fibrosis (scored according to revised Banff 1997 criteria) in consecutive protocol biopsies | 24 months post-transplantation

SECONDARY OUTCOMES:
Graft function (eGFR, calculated with the Modification of Diet in Renal Disease formula) | 24 months post-transplantation
Proteinuria (measured as g/g creatinine in a 24-hr urine collection) | 24 months post-transplantation
Urinary CTGF concentration | 24 months post-transplantation
Intra-graft expression of CTGF | 24 months post-transplantation
Urinary markers of tubular injury and dysfunction | 24 months post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Kuypers, MD, PhD, Principal Investigator — Laboratory of Nephrology, University Hospitals Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium